CLINICAL TRIAL: NCT03110744
Title: CDK4/6 Inhibition in Locally Advanced/Metastatic Chordoma (NCT-PMO-1601)
Brief Title: CDK4/6 Inhibition in Locally Advanced/Metastatic Chordoma
Acronym: NCT-PMO-1601
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard F Schlenk, Prof. Dr. med. Richard F. Schlenk (Coordinating Investigator), University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2016-415 / Chordoma
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Chordoma
MeSH Terms: conditions — Chordoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib (Experimental): application on 21 consecutive days of a 28 days cycle
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — application on 21 consecutive days of a 28 days cycle
  Other Names: Ibrance

SUMMARY:
In chordoma cell lines and patient biopsies, the p16 (CDKN2A) tumor suppressor is consistently deleted. Thus, chordomas are an example of a tumor with universal activation of the cyclin-dependent kinases 4 and 6 (CDK4/6) pathway, and experiments with patient-derived chordoma cell lines demonstrate aberrant CDK4/6 activity downstream of p16 loss can be efficiently inhibited by the CDK4/6 inhibitor palbociclib, resulting in reduced proliferation and growth of neoplastic cells. The investigators aim to conduct a phase II clinical trial to evaluate the efficacy of the small-molecule CDK4/6 inhibitor palbociclib in patients with locally advanced/metastatic chordoma who are not candidates for standard therapy. The primary objective is disease control in patients with chordoma treated with palbociclib as single agent. The study design of this phase II study is based on a Simon two-stage design.

DETAILED DESCRIPTION:
Chordoma is a rare bone tumor with slow growth. The standard treatment is en bloc excision, but the site of origin of the disease often prevents complete surgery. For these patients, debulking surgery followed by radiation therapy (RT) or high-dose RT alone can be an alternative. However, local relapses or more rarely metastatic disease frequently occur, and there is no efficient standard systemic therapy available. Only very limited responses are seen with chemotherapy or targeted agents, such as imatinib and lapatinib. In chordoma cell lines and patient biopsies, the p16 (CDKN2A) tumor suppressor is consistently deleted. Thus, chordomas are an example of a tumor with universal activation of the CDK4/6 pathway, and experiments with patient-derived chordoma cell lines demonstrate aberrant CDK4/6 activity downstream of p16 loss can be efficiently inhibited by the CDK4/6 inhibitor palbociclib, resulting in reduced proliferation and growth of neoplastic cells. The investigators aim to conduct a phase II clinical trial to evaluate the efficacy of the small-molecule CDK4/6 inhibitor palbociclib in patients with locally advanced/metastatic chordoma who are not candidates for standard therapy. The primary objective is disease control in patients with chordoma treated with palbociclib as single agent. The study design of this phase II study is based on a Simon two-stage design. This trial will establish whether the overreliance of chordomas on the activation of the CDK4/6-Retinoblastoma 1 (RB1) pathway can be exploited for therapeutic benefit. Based on previous experience with 125 mg palbociclib once daily for 21 days followed by 7 days of rest in patients with breast cancer, liposarcoma, non-small cell lung cancer, hepatocellular carcinoma, ovarian cancer, mantle-cell lymphoma, and glioblastoma, this regimen is chosen. Based on a Simons optimal two-stage design the disease control rate (DCR) will be the primary end-point, whereby response is defined as complete response (CR), partial response (PR), or stable disease (SD) according to RECIST v1.1 criteria after six cycles. For sample size calculation the investigators estimate a poor response with 10% and a good response with 25% (power, 80%; alpha, 5%) leading to a first stage of 18 patients and, if three or more patients responded to a second stage with additional 25 patients (total n=43).

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic chordoma with confirmed diagnosis in a reference pathology (with immunohistology for epithelial membrane antigen, S100, Brachyury, Integrase interactor 1 (INI-1)) not amenable to curative treatment with surgery or radiotherapy
* At least one measurable tumor lesion according to RECIST 1.1 criteria
* Loss of p16 determined immunohistochemically or CDKN2A/B genomically, presence of CDK4/6 and RB1 determined immunohistochemically or by RNA-Sequencing.
* Age ≥ 18 years, no upper age limit
* Availability of tissue blocks preferably not older than 12 months for immunohistologic assessment (if no adequate material is available, re-biopsy should be considered before entering the study)
* No chemotherapy two weeks before study
* Non-pregnant and non-nursing. Women of child-bearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 72 hours prior to registration (WOCBP is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 months).
* Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (double barrier contraceptive method (IUD, condome), tubal ligation, or partner's vasectomy) while on therapy and for 14 weeks after the last dose of therapy. Hormonal contraception alone is an inadequate method of birth control. Female patients must agree not to donate lactation during treatment and until 14 weeks after end of treatment.
* Men must agree not to father a child and must use a latex condom during any sexual contact with WOCBP while receiving therapy and for 14 weeks after therapy is stopped, even if they have undergone successful vasectomy. Sperm donation is not permitted for the same time interval.
* Signed written informed consent
* Performance status ≤ 2 according to Eastern Cooperative Oncology Group (ECOG) /World Health Organization (WHO) criteria
* Ability of patient to understand the character and individual consequences of clinical trial

Exclusion Criteria:

* Prior treatment with palbociclib or known intolerance/allergy to the compound or any ingredient (acquired or hereditary).
* Prior treatment with other CDK4/6 inhibitors
* Co-therapy with strong/potent CYP3A inducers and/or inhibitors, (e.g., Clarithromycin, Indinavir, Itraconazol, Ketoconazol, Lopinavir/Ritonavir, Nefazodon, Nelfinavir, Posaconazol, Saquinavir, Telaprevir, Telithromycin, Voriconazol, and St. John's Wort [Hypericum perforatum])) while on treatment with study drug.
* Co-therapy with corticosteroids above 7.5 mg prednisolone/prednisone equivalent
* Anticancer treatment less than 2 weeks prior to study treatment
* Organ insufficiency: creatinine clearance <30ml/min; total bilirubin > 1.5x upper normal serum level; AST > upper normal serum level ; abnormal blood counts; heart failure (New York Heart Association (NYHA) III/IV); uncontrolled hypertension; unstable angina; serious cardiac arrhythmia; severe obstructive or restrictive ventilation disorder
* Clinical signs of active infection (° grade 2-CTCAE Vers.5.0)
* Patients with a "currently active" second malignancy other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if the patients have completed therapy and are considered by the patients physician to be at less than 30% risk of relapse within one year.
* Severe neurologic or psychiatric disorder interfering with ability of giving informed consent
* Known or suspected active alcohol or drug abuse
* Known positivity for HIV, active hepatitis A virus (HAV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection
* Uncontrolled central nervous system (CNS) involvement (treatment for CNS-involvement prior to inclusion is allowed)
* Cytopenia: platelets <100 G/l, neutrophils <1.0 G/l, hemoglobin <10.0 g/dl
* corrected QT interval (QTc) >470 msec (based on the mean value of triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome, or known history of QTc prolongation or Torsade de Pointes
* Uncontrolled electrolyte disorders that can aggravate the effects of a QTc-prolonging drug (e.g., hypocalcemia, hypokalemia, hypomagnesemia)
* Participation in other ongoing interventional clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 6 months
  The primary endpoint is the DCR after six cycles of palbociclib, which is defined as the presence of at least one confirmed complete response (CR) or confirmed partial response (PR) or stable disease (SD) according to RECIST version 1.1.

SECONDARY OUTCOMES:
Tumor response rate (TRR) | 6 months
  • defined as the sum of complete remission (CR) and partial remission (PR) according to RECIST version 1.1 after six cycles of study medication.
Progression-free survival (PFS) | 6 months
  • defined as the time from first administration of the Investigational Medicinal Product (IMP) to radiologically confirmed progression of disease or death from any cause, whichever occurs first. Patients without the event are censored on the last date of follow-up.
Overall survival (OS) | 6 months
  • defined as the time from first administration of the IMP to time of death from any cause. Patients without the event are censored on the last date of follow-up.
Safety (toxicity, tolerability): Toxic effects will be graded according to CTCAE v4.03. | 6 months
  • Toxic effects will be graded according to CTCAE v4.03.
Quality of life (QoL) | 6 months
  • QoL will be assessed by the EORTC Quality of Life Core Questionnaire (QLQ-C30), supplemented by information on self-assessed concomitant diseases and demographics initially, after the first, and after the sixth 28-day treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Fröhling, Prof. Dr., Principal Investigator — NCT Heidelberg
Locations (3):
- Germany (3):
  - Universitätsklinikum Essen, Essen
  - National Center for Tumor Diseases, Heidelberg
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT03110744/Prot_001.pdf